CLINICAL TRIAL: NCT07286656
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Subcutaneous Dose of GenSci098 in Patients With Graves' Disease
Brief Title: A Study of GensSci098 in Subjects With Graves' Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GenSci098-102
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Safety; Tolerability; GenSci098; Graves Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GenSci098 (Experimental)
  Interventions: Drug: GenSci098

INTERVENTIONS:
Drug: GenSci098 — * Administration: Only one dose of GenSci098 will be given.
  * Route of Administration: Subcutaneous (injected under the skin).
  * Dose Levels: • Dose 1 • Dose 2• Dose 3• Dose 4

SUMMARY:
To evaluate the safety and tolerability of single ascending subcutaneous doses of GenSci098 in patients with Graves' Disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Voluntary signed informed consent.
* Confirmed diagnosis of diffuse toxic goiter (Graves' disease).
* Abnormal thyroid function tests (e.g., elevated T3, T4, and suppressed TSH).
* No prior or recent use of antithyroid medications (discontinued for at least 4 weeks).
* No thyroid eye disease or only mild thyroid eye disease.
* Female participants must be postmenopausal, surgically sterile, or using a highly effective method of contraception.
* Male participants must agree to practice abstinence, use a highly effective method of contraception， or have undergone vasectomy.
* Ability to comply with the follow-up schedule and understand and adhere to the study requirements.

Exclusion Criteria:

* Non-diffuse toxic goiter-induced hyperthyroidism.
* Previous radioactive iodine treatment or thyroid surgery.
* History or risk of thyroid storm.
* Use of thyroid hormone medications within the past 6 weeks.
* Thyroid eye disease treated with radiation/surgery,or need for urgent surgery.
* Optic nerve lesions or corneal damage.
* Use of steroids or immunosuppressants within the past 3 months.
* Inability to quit smoking during the study.
* Allergy to the study drug or monoclonal antibodies.
* Participation in another clinical trial within the past 3 months.
* Abnormal electrocardiogram.
* Significant hepatic or renal dysfunction.
* Pregnancy,breastfeeding,or positive pregnancy test.
* Positive for HIV,syphilis,hepatitis B,or hepatitis C.
* History of drug or substance abuse.
* Other autoimmune diseases requiring treatment.
* History of malignant tumors.
* Splenectomy or major surgery within the past 6 months.
* Severe cardiovascular,pulmonary,hepatic,renal,neurological,or hematological diseases.
* Other conditions deemed unsuitable by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-11-19 (Estimated); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) (physical examination, vital signs, laboratory tests, 12-lead electrocardiogram [ECG]). | 141 days
  This outcome measure assesses the incidence and severity of adverse events (AEs) experienced by participants during the study. AEs will be monitored through physical examinations, vital signs, laboratory tests, and 12-lead electrocardiograms (ECGs). The assessment period spans from the first dose of the study intervention to 141 days post-dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyan Shan, PHD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China